CLINICAL TRIAL: NCT04228211
Title: Utrecht Prostate Cohort for Cancer Treatment Intervention Studies and Long-term Evaluation
Acronym: UPC
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Professor of epidmiology, UMC Utrecht
Other Study IDs: NL70198.041.19
Record Dates: First submitted 2020-01-03; First posted 2020-01-14 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; trials within cohorts (TwiCs) design
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Rationale: Prostate cancer is the most common cancer in men worldwide. Survival rates are high due to the typically non-aggressive nature of disease and effective treatments. Radical treatments such as surgery and radiotherapy often cause toxicity and long term side effects. Based on current available literature, the choice for primary therapy for clinically localised prostate cancer has a negative impact on cancer-specific quality of life (QOL). New interventional treatments are being developed. The investigators aim to build a multidisciplinary prostate cancer cohort which will serve as a multi-trial facility for interventional treatment studies. The Trials within Cohorts (TwiCs) design, also known as cohort multiple Randomized Controlled Trial design (cmRCT) will be conducted and as a prospective registry for assessment of long-term safety, performance and effectiveness new treatment interventions.

Objective: To set up a cohort that will serve as a multi-trial platform and facilitate evaluation of new interventional treatment for prostate cancer.

Study design: Observational, prospective cohort study, according to the 'Trials within Cohorts' (TwiCs) design.

Study population: All patients with newly diagnosed histologically proven prostate cancer.

Main study parameters/endpoints: Clinical parameters (e.g. co-morbidity, oncological history, symptoms, imaging, technical and treatment data), clinical endpoints (e.g. toxicity, and survival outcomes) and patient reported outcomes (e.g. QOL).

DETAILED DESCRIPTION:
Introduction to Trials within Cohorts (TwiCs) design:

With "Utrecht Prostate Cohort for cancer treatment intervention studies and long term evaluation"(UPC) the investigators aim to: (1) develop an ongoing observational database with short- and long-term clinical and patient-reported outcomes during and after treatment for newly diagnosed prostate cancer. (2) Provide a cohort for multiple randomized controlled trials for evaluation of new treatment interventions for prostate cancer. The initial collaborating centers in the UPC study are the University Medical Center (UMC) Utrecht and the St. Antonius Hospital Nieuwegein both regional tertiary referral centers, covering the total spectrum of prostate cancer care. All patients with newly diagnosed histologically proven prostate cancer presenting at the UMC Utrecht or the St. Antonius Hospital Nieuwegein are eligible for participation in UPC.

The investigators will implement a cohort-based trial infrastructure following the TwiCs design. The TwiCs design is an efficient alternative to the classic randomized controlled trial (RCT) and is considered particularly suitable for evaluation of image guided interventions. In TwiCs, prospective cohorts or registries serve as facilities for simultaneous and randomised evaluation of multiple interventions for the same condition. The basis of the TwiCs is a large prospective observational cohort of patients with the condition of interest (e.g. prostate cancer), who (in principle) undergo standard treatment and for whom relevant short and long term outcome measures are captured. For each new intervention, all eligible patients within the cohort are identified. Some of these eligible patients will be randomly selected and offered the new intervention. The outcomes of these randomly selected patients are then compared to those of the eligible patients receiving usual care. The same process can be repeated (simultaneously) for other experimental interventions. Advantages of the TwiCs are its ability to facilitate multiple randomised evaluations, the improved comparability between trials and the patient-centred informed consent procedure. Higher numbers of eligible patients are expected to be enrolled in studies, improving generalisability of results. Also, the cohorts can serve as patient pools from which patients can be selected for the R-IDEAL (Radiotherapy-Idea, Development, Exploration, Assessment, and Long-term evaluation) stage 2a technical development studies, and as registries for long term follow-up studies.

In the Utrecht region, the investigators have set up multiple cohorts according to the TwiCs design, in which over 4000 patients have been enrolled, and in which four trials and dozens of technical development and observational studies are running.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with newly diagnosed histologically proven prostate cancer, referred for radiation treatment to the Radiotherapy Department of the UMC Utrecht or for prostatectomy, watchful waiting or active surveillance to the Urology Department of St. Antonius hospital or the Urology Department of the UMC Utrecht.
* Informed consent - at least - for use of routinely collected clinical data and to fill out questionnaires.

Exclusion Criteria:

* Mentally incompetent patients.
* Inability to understand the Dutch language.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosed histologically proven prostate cancer, referred for radiation treatment to the Radiotherapy Department of the UMC Utrecht or for prostatectomy, watchful waiting or active surveillance to the Urology Department of St. Antonius hospital or the Urology Department of the UMC Utrecht will be eligible to be enrolled in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-02-05 (Estimated); Study Completion 2033-02-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Quality of Life | Up to 10 years after treatment
  Assesment of Health-related quality of life in prostate cancer patients undergoing treatment
Occurence of toxicity (adverse events) | Up to 10 years after treatment
  All toxicity occurring during or after treatment will be registered according to the Common Terminology Criteria for Adverse Events (CTCAE version 5) and Clavien Dindo classification, for radiotherapy and surgery respectively.
Occurence of disease recurrence/progression | Up to 10 years after treatment
  Biochemical prostate specifice antigen (PSA) recurrence/progression and recurrence/progression based on medical imaging

SECONDARY OUTCOMES:
Survival | Up to 10 years after treatment
  Survival of participating patients will be recorded using the follow up questionnaires (returned by family members) or are derived from the Municipal Personal Records Database (in Dutch: Gemeentelijke Basisadministratie, GBA).

CONTACTS AND LOCATIONS:
Overall Officials: Helena M. Verkooijen, MD, PhD, Principal Investigator — UMC Utrecht; Jochem R.N. van der Voort van Zyp, MD, PhD, Principal Investigator — UMC Utrecht; Harm H.E. van Melick, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Study protocol will be submitted for publication in a peer reviewed (international) scientific journal

REFERENCES:
- [Derived] Teunissen FR, Willigenburg T, Meijer RP, van Melick HHE, Verkooijen HM, van der Voort van Zyp JRN. The first patient-reported outcomes from the Utrecht Prostate Cohort (UPC): the first platform facilitating 'trials within cohorts' (TwiCs) for the evaluation of interventions for prostate cancer. World J Urol. 2022 Sep;40(9):2205-2212. doi: 10.1007/s00345-022-04092-2. Epub 2022 Jul 21. PMID 35861861